CLINICAL TRIAL: NCT05165654
Title: Improving Hallucinations by Targeting the Right Superior Temporal Sulcus With Electrical Stimulation
Brief Title: Improving Hallucinations by Targeting the rSTS With tES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Paulo Lizano, Assistant Professor, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P001016X
Record Dates: First submitted 2021-11-17; First posted 2021-12-21 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Hallucinations, Auditory; Psychosis
Keywords: Transcranial Electrical Stimulation; Electroencephalography
MeSH Terms: conditions — Hallucinations; Psychotic Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active Stimulation with TDCS (Experimental): 10 tDCS; Two, twenty-minute sessions of tDCS to the rSTS for 5 days (10 total sessions).
  Interventions: Device: Transcranial Electrical Stimulation
- SHAM Stimulation (Sham Comparator): 10 passive sham control; Two, twenty-minute sessions of passive sham control to the rSTS for a 30 second ramped up and down at the beginning and end of the 20 min period for 5 days (10 total sessions).
  Interventions: Device: Transcranial Electrical Stimulation

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — Transcranial electrical stimulation

SUMMARY:
Hallucinations are a core diagnostic feature of psychotic disorders. They involve different sensory modalities, including auditory, visual, olfactory, tactile, and gustatory hallucinations, among others. Hallucinations occur in multiple different neurological and psychiatric illnesses and can be refractory to existing treatments. Auditory hallucinations and visual hallucinations are found across diagnostic categories of psychotic disorders (schizophrenia, schizoaffective, bipolar disorder). Despite visual hallucinations being approximately half as frequent as auditory hallucinations, they almost always co-occur with auditory hallucinations, and are linked to a more severe psychopathological profile. Auditory and visual hallucinations at baseline also predict higher disability, risk of relapse and duration of psychosis after 1 and 2 years, especially when they occur in combination. Using a newly validated technique termed lesion network mapping, researchers demonstrated that focal brain lesions connected to the right superior temporal sulcus (rSTS) plays a causal role in the development of hallucinations. The rSTS receives convergent somatosensory, auditory, and visual inputs, and is regarded as a site for multimodal sensory integration. Here the investigators aim to answer the question whether noninvasive brain stimulation when optimally targeted to the rSTS can improve brain activity, sensory integration, and hallucinations.

DETAILED DESCRIPTION:
Functional neuroimaging studies have identified neural correlates of hallucinations across multiple brain regions. Some studies suggest a common neuroanatomical substrate independent of the sensory modality, while others suggest different neural correlates for different types of hallucinations. However, whether these neuroimaging findings represented a cause, consequence or epiphenomenon of hallucinations was unclear until recently. Using lesion network mapping, researchers demonstrated that focal brain lesions play a causal role in the development of hallucinations and can occur in different brain locations, both inside and outside sensory pathway, and that greater than 90% of lesion locations causing hallucinations are negatively connected to the right superior temporal sulcus (rSTS). The rSTS is known to play a role in social cognition, biological motion, audiovisual integration, and speech. Hence, when spontaneous activity decreases at lesion locations causing hallucinations, spontaneous activity in the rSTS increases, the exact pattern thought to predispose to hallucinations. Additionally, functional connectivity within this region is abnormal in patients with visual and auditory hallucinations. Therefore, the association between rSTS connectivity and hallucinations would suggest this region may be optimal for modulation via non-invasive brain stimulation.

One method by which cortical excitability can be altered is with transcranial direct current stimulation (tDCS), a non-invasive brain stimulation technique. High definition tDCS (HD-tDCS) is a refined version of tDCS with improved spatial precision of cortical stimulation. This involves the application of a weak electrical current (1-2 mA) delivered to the brain via scalp electrodes. tDCS can modulate cortical excitability, where anodal stimulation tends to increase (i.e. the resting potential becomes less negative) and cathodal stimulation tends to decrease the underlying membrane potential (i.e. the resting potential becomes more negative). While tDCS is a promising adjunctive treatment of auditory hallucinations and negative symptoms in schizophrenia, less is known about its role in treating hallucinations overall. To date, no study has non-invasively stimulated the rSTS with tDCS in psychosis and examined its effects on hallucinations. However, there are studies in healthy volunteers showing that anodal stimulation to the STS resulted in increased auditory false perceptions, while cathodal stimulation decreased false perceptions and was lower than the sham condition. Taken together, the recent lesion network mapping identifying the rSTS as a major source of hallucinations combined with prior studies showing that the rSTS is associated with hallucinations suggest that it may be possible to alleviate hallucinations by designing a tDCS protocol that targets the rSTS with cathodal stimulation. Technological advances in noninvasive neuromodulation and electrical field modeling further allow us to create a tDCS protocol specifically guided by the results of lesion network mapping studies with high spatial resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-50 years of age
2. Proficient in English
3. Able to give informed consent
4. Actively experiencing hallucinations (tactile, auditory, visual, etc.)
5. Has not recently participated in tES/TMS treatments

Exclusion Criteria:

1. Substance abuse or dependence (w/in past 6 months)
2. Those who are pregnant/breastfeeding
3. History of head injury with > 15 minutes of loss of consciousness/mal sequelae
4. DSM-V intellectual disability
5. Having a non-removable ferromagnetic metal within the body (particularly in the head)
6. History of seizures

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-06-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Lizano, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through patient conversations and advertisements.
Pre-assignment Details: Individuals performed a full clinical assessment including a structured clinical interview and medical history review to confirm diagnosis. Individuals were required to have a history or current hallucinations (visual, auditory, tactile, etc.) to participate in the study. Participants were then randomized to one of the two arms of the study (active tDCS or sham) targeting the right superior temporal sulcus.
Groups:
- Active Stimulation With TDCS: tDCS; Two, twenty-minute sessions of tDCS to the rSTS for 5 days (10 total sessions).
  Transcranial Electrical Stimulation: Transcranial electrical stimulation
- SHAM Stimulation: Passive sham control; Two, twenty-minute sessions of passive sham control to the rSTS for a 30 second ramped up and down at the beginning and end of the 20 min period for 5 days (10 total sessions).
  Transcranial Electrical Stimulation: Transcranial electrical stimulation
Period: Overall Study
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Started | 6 | 6
Baseline | 6 | 6
Day 5 | 6 | 6
1 Month | 5 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.7 (8.3) | 37.5 (14.8) | 37.1 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 5 | 6 | 11
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Prior/Current Hallucinations [Count of Participants; unit: Participants] | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: Measuring total psychosis symptoms score (Total score minimum = 30, maximum = 210); General symptoms (minimum score = 16, maximum score = 112); Negative Symptoms (minimum score = 16, maximum score = 112); and Positive Symptoms (minimum score = 16, maximum score = 112); higher scores represent higher severity of symptoms
Time Frame: Change from baseline to day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 60.5 [47.75 to 77] | 60 [53.75 to 69.25]
  Day 5 | 56 [44.25 to 75.25] | 63 [59 to 70]

2. Primary Outcome: Positive and Negative Syndrome Scale (PANSS)
Description: as for outcome 1
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation on 1 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 60.5 [47.75 to 77] | 60 [53.75 to 69.25]
  1 Month | 58.5 [47 to 67.75] | 70.5 [60.25 to 83.75]

3. Primary Outcome: University of Miami Parkinson's Disease Hallucinations Questionnaire (UM-PDHQ)
Description: Measuring severity and duration of hallucinations; 20-item questionnaire to be used as a screening instrument to assess hallucinations (6 quantitative and 14 qualitative items); higher scores represent higher severity of symptoms. Total quantitative score (min = 0; max = 14).
Time Frame: Change from baseline to day 5
Population: Total quantitative score reported (min = 0; max = 14)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 1.85 [1.725 to 2.025] | 1.9 [1.85 to 2.0125]
  Day 5 | 1.3 [1.25 to 1.35] | 2 [1.8 to 2.2]

4. Primary Outcome: University of Miami Parkinson's Disease Hallucinations Questionnaire (UM-PDHQ)
Description: as for outcome 3
Time Frame: Change from baseline to month follow-up
Population: Total quantitative score reported (min = 0; max = 14)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 1.85 [1.725 to 2.025] | 1.9 [1.85 to 2.0125]
  1 Month | 1.4 [1.05 to 1.6875] | 2.35 [2.05 to 2.4]

5. Primary Outcome: 7-item Auditory Hallucinations Rating Scale (AHRS)
Description: Measuring severity and duration of hallucinations; severity for each item is rated on a 7-point scale; higher scores represent higher severity of symptoms. Total score (0-41).
Time Frame: Change from baseline to day 5
Population: Total score reported (0-41).
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 0 [0 to 0] | 8 [0 to 19.75]
  Day 5 | 0 [0 to 0] | 6 [0 to 22.5]

6. Primary Outcome: 7-item Auditory Hallucinations Rating Scale (AHRS)
Description: as for outcome 5
Time Frame: Change from baseline to month follow-up
Population: Total score reported (0-41)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 0 [0 to 0] | 8 [0 to 19.75]
  1 Month | 0 [0 to 0] | 6 [0 to 23.25]

7. Secondary Outcome: Auditory Steady State Evoked Potential
Description: Raw data was cleaned for artifacts (excessive noise) and segmented in cleaned epochs based on stimulus onset. Post preprocessing stages, the signal reported was derived from using a time-frequency transformation and analysis, which is conceptualized as oscillatory power in decibels (10*log10) at a particular auditory frequency of interest.
Time Frame: Change from baseline to day 5
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Mean (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | 0.369044853 [0.091708253 to 0.624277228] | 0.434681797 [0.16328823 to 0.643059721]
  Day | 0.259385513 [0.190658708 to 0.314372544] | 0.257550439 [-0.046862077 to 0.352363789]

8. Secondary Outcome: Auditory Steady State Evoked Potential
Description: as for outcome 7
Time Frame: Change from baseline to month follow-up
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Median (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | 0.369044853 [0.091708253 to 0.624277228] | 0.434681797 [0.16328823 to 0.643059721]
  1 Month | 0.307252913 [0.241709825 to 0.677070695] | 0.221649958 [-0.021732331 to 0.406676752]

9. Secondary Outcome: Steady State Visual Evoked Potential
Description: Raw data was cleaned for artifacts (excessive noise) and segmented in cleaned epochs based on stimulus onset. Post preprocessing stages, the signal reported was derived from using a time-frequency transformation and analysis, which is conceptualized as oscillatory power in decibels (10*log10) at a particular visual frequency of interest.
Time Frame: Change from baseline to day 5
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Median (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | -0.62131125 [-0.726391384 to -0.074934424] | -0.046333327 [-0.103732736 to 0.052670088]
  Day 5 | -0.101487523 [-0.548558447 to 0.099856615] | -0.061733608 [-0.291644849 to 0.143966164]

10. Secondary Outcome: Steady State Visual Evoked Potential
Description: as for outcome 9
Time Frame: Change from baseline to month follow-up
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Median (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | -0.62131125 [-0.726391384 to -0.074934424] | -0.046333327 [-0.103732736 to 0.052670088]
  1 Month | 0.276320034 [0.09372428 to 0.34434154] | -0.342125912 [-0.525993493 to -0.203782791]

11. Secondary Outcome: Cross Modal Steady State Evoked Potential
Description: Raw data was cleaned for artifacts (excessive noise) and segmented in cleaned epochs based on stimulus onset. Post preprocessing stages, the signal reported was derived from using a time-frequency transformation and analysis, which is conceptualized as oscillatory power in decibels (10*log10) at a particular visual/auditory frequency of interest.
Time Frame: Change from baseline to day 5
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Median (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | -0.129873057 [-0.351085988 to -0.039036888] | -0.225582699 [-0.369160721 to -0.084290267]
  Day 5 | -0.227227968 [-0.314087578 to -0.209605677] | -0.309958523 [-0.479995017 to -0.140836317]

12. Secondary Outcome: Cross Modal Steady State Evoked Potential
Description: as for outcome 11
Time Frame: Change from baseline to month follow-up
Population: 1 individual in the active TDCS group had unusable data due to poor data quality.
Measure: Median (Inter-Quartile Range); unit: decibels
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 5 | 6
decibels
  Baseline | -0.129873057 [-0.351085988 to -0.039036888] | -0.225582699 [-0.369160721 to -0.084290267]
  1 Month | -0.372064254 [-0.395091449 to -0.264603929] | -0.370288832 [-0.480430263 to -0.146267599]

13. Secondary Outcome: Resting State EEG
Description: Measuring neural activity at rest consisting of 5 minutes of eyes-open resting-state EEG (rsEEG) was recorded. Fast Fourier transformations were conducted on data, resulting in 4 frequency bands: delta/theta, alpha, beta, and gamma.
Time Frame: Change from baseline to 5 day
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
microvolts
  Baseline Delta/Theta Range (1-8hz) | -6.067479336 [-8.358364857 to -5.444418054] | -9.836502863 [-10.87640284 to -6.060701682]
  Day 5 Delta/Theta Range (1-8hz) | -6.538377742 [-8.949555683 to -5.160262915] | -8.837371992 [-11.64394669 to -7.549197399]
  Baseline Alpha (8-12hz) | -7.920960953 [-10.83320875 to -7.295414497] | -11.66579035 [-13.69578824 to -7.820418988]
  Day 5 Alpha (8-12hz) | -7.433306198 [-10.21438969 to -7.043908117] | -10.07675116 [-13.61574437 to -7.162213165]
  Baseline Beta (13-30hz) | -15.99107017 [-16.44864468 to -15.41891723] | -17.88706322 [-18.60085714 to -16.64276514]
  Day 5 Beta (13-30hz) | -15.97882887 [-16.30148928 to -15.67218914] | -17.45169236 [-17.80617123 to -15.82596502]
  Baseline Gamma (30-55hz) | -22.64365385 [-23.36454231 to -21.38378251] | -22.02556837 [-24.09400191 to -20.51039388]
  Day 5 Gamma (30-55hz) | -23.79503055 [-24.38033537 to -20.99613743] | -22.638985 [-23.25493645 to -21.12844812]

14. Secondary Outcome: Resting State EEG
Description: as for outcome 13
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation of 1 Month data
Measure: Median (Inter-Quartile Range); unit: microvolts
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
microvolts
  Baseline Delta/Theta Range (1-8hz) | -6.067479336 [-8.358364857 to -5.444418054] | -9.836502863 [-10.87640284 to -6.060701682]
  1 Month Delta/Theta Range (1-8hz) | -5.891239776 [-7.30798828 to -4.582039071] | -8.925939219 [-10.09990467 to -7.862654867]
  Baseline Alpha (8-12hz) | -7.920960953 [-10.83320875 to -7.295414497] | -11.66579035 [-13.69578824 to -7.820418988]
  1 Month Alpha (8-12hz) | -9.390036281 [-10.94620211 to -8.24923518] | -7.367402407 [-9.002447243 to -7.084971382]
  Baseline Beta (12-30hz) | -15.99107017 [-16.44864468 to -15.41891723] | -17.88706322 [-18.60085714 to -16.64276514]
  1 Month Beta (13-30hz) | -16.0281252 [-17.60044849 to -15.79720705] | -16.27626797 [-18.23084259 to -15.95296812]
  Baseline Gamma (30-55hz) | -22.64365385 [-23.36454231 to -21.38378251] | -22.02556837 [-24.09400191 to -20.51039388]
  1 Month Gamma (30-55hz) | -23.89591029 [-24.94829518 to -22.12361733] | -22.95515728 [-24.30097235 to -22.21405322]

15. Secondary Outcome: Biological Motion
Description: Measuring the percent correct of detected motion by presenting a simulated walker; difficulty is increased by the level of random noise around stimuli. 20 trials are presented. Higher scores (0-100%) indicate a better ability to detect motion.
Time Frame: Change from baseline to 5 day
Measure: Median (Inter-Quartile Range); unit: percentage correct
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
percentage correct
  Baseline | 87.5 [76.25 to 98.75] | 85 [61.25 to 93.75]
  Day 5 | 95 [87.5 to 98.75] | 72.5 [51.25 to 93.75]

16. Secondary Outcome: Biological Motion
Description: as for outcome 15
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation of 1 Month data
Measure: Median (Inter-Quartile Range); unit: percentage correct
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
percentage correct
  Baseline | 87.5 [76.25 to 98.75] | 85 [61.25 to 93.75]
  1 Month | 95 [87.5 to 95] | 85 [67.5 to 95]

17. Secondary Outcome: Neurological Evaluation Scale; Sensory Integration
Description: Measuring the percent correct of auditory and visual integration; auditory stimuli partners are matched to visual stimuli; difficulty is increased with more complex patterns
Time Frame: Change from baseline to 5 day
Population: Data was unable to be obtained for due to the a technique problem in code for the task that resulted in incorrectly quantifying outcomes.
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 0 | 0

18. Secondary Outcome: Neurological Evaluation Scale; Sensory Integration
Description: as for outcome 17
Time Frame: Change from baseline to month follow-up
Population: as for outcome 17
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 0 | 0

19. Secondary Outcome: Global Assessment of Function (GAF)
Description: Measuring global functioning; severity of symptoms related to day-to-day life on a scale of 0 to 100; higher scores represent higher severity of symptoms
Time Frame: Change from baseline to day 5
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 60.5 [53.25 to 64] | 57.5 [43.75 to 60]
  Day 5 | 60.5 [52.5 to 67.75] | 53 [42.75 to 58.75]

20. Secondary Outcome: Global Assessment of Function (GAF)
Description: as for outcome 19
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation on 1 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 60.5 [53.25 to 64] | 57.5 [43.75 to 60]
  1 Month | 61.5 [56.25 to 68.25] | 54 [51.5 to 59.5]

21. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: Measuring total depression scores; 10 item scale related to depressive episodes (total score 0-60); higher scores represent higher severity of symptoms
Time Frame: Change from baseline to 5 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 7 [3.5 to 16.5] | 7.5 [4.75 to 10.25]
  Day 5 | 6 [2.5 to 18.5] | 13.5 [5.5 to 20]

22. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: as for outcome 21
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation on 1 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 7 [3.5 to 16.5] | 7.5 [4.75 to 10.25]
  1 Month | 5.5 [4.25 to 19.5] | 13 [10.5 to 15.5]

23. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: Measuring total Mania scores; 11 items used to access severity of mania (total score 0-60); higher scores represent higher severity of symptoms
Time Frame: Change from baseline to 5 day
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 2.25 [0.625 to 14] | 7 [3.625 to 11.875]
  Day 5 | 1.25 [0.125 to 11.375] | 14 [6.375 to 14.875]

24. Secondary Outcome: Young Mania Rating Scale (YMRS)
Description: as for outcome 23
Time Frame: Change from baseline to month follow-up
Population: 'Mice" R package used for multiple imputation on 1 Month data
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 2.25 [0.625 to 14] | 7 [3.625 to 11.875]
  1 Month | 2 [1.25 to 10.25] | 8.75 [5.25 to 14.875]

25. Secondary Outcome: Brief Assessment of Cognition (BACS)
Description: Measuring cognition; cognitive domains assessed include memory, working memory, processing speed, executive functions and verbal fluency. Higher scores indicate greater cognitive ability on a given task.
Time Frame: Change from baseline to 5 day
Population: BACS total score reported. Summed from all subcategories of cognition (memory, working memory, processing speed, executive function and verbal fluency scores). Scores transformed into Z scores based off standardized transformations provided by the test makers. 0 represents the population mean for healthy controls. Standard deviations above the mean represent better cognitive ability.
Measure: Median (Inter-Quartile Range); unit: z score on test
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
z score on test
  Baseline | 0.58 [-0.7075 to 1.005] | -0.8 [-1.5325 to -0.4275]
  Day 5 | -0.15 [-1.355 to 0.5375] | -1.065 [-1.7775 to -0.5475]

26. Secondary Outcome: Brief Assessment of Cognition (BACS)
Description: as for outcome 25
Time Frame: Change from baseline to month follow-up
Population: 'Mice" R package used for multiple imputation on 1 Month data; BACS total score reported. BACS total score reported. Summed from all subcategories of cognition (memory, working memory, processing speed, executive function and verbal fluency scores). Scores transformed into Z scores based off standardized transformations provided by the test makers. 0 represents the population mean for healthy controls. Standard deviations above the mean represent better cognitive ability.
Measure: Median (Inter-Quartile Range); unit: z score on test
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
z score on test
  Baseline | 0.58 [-0.7075 to 1.005] | -0.8 [-1.5325 to -0.4275]
  1 Month | -0.07 [-0.5775 to 0.7525] | -1.425 [-1.825 to -0.8225]

27. Secondary Outcome: Symptom Checklist-90
Description: Measuring total psychiatric symptoms; 90 symptoms and evaluates nine symptomatic dimensions; higher scores represent higher severity of symptoms. Total score range 0 to 360
Time Frame: Change from baseline to 5 day
Population: Total score assesses psychological distress through 90 items reported. Total score reported, range 0 to 360.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 56.5 [21.75 to 119.75] | 81.5 [56.5 to 95.25]
  Day 5 | 33 [9.25 to 56] | 84.5 [69.25 to 95.25]

28. Secondary Outcome: Symptom Checklist-90
Description: Measuring total psychiatric symptoms; 90 symptoms and evaluates nine symptomatic dimensions; higher scores represent higher severity of symptoms.Total score range 0 to 360.
Time Frame: Change from baseline to month follow-up
Population: 'Mice' R package used for multiple imputation on missing data. Total score assesses psychological distress through 90 items reported. Total score reported, range 0 to 360.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
Number analyzed (Participants) | 6 | 6
score on a scale
  Baseline | 56.5 [21.75 to 119.75] | 81.5 [56.5 to 95.25]
  1 Month | 42 [16.5 to 102] | 95.5 [79.5 to 124.25]

ADVERSE EVENTS:
Time Frame: Up to 1 month period after study participation
Arm/Group | Active Stimulation With TDCS | SHAM Stimulation
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation With TDCS (N=6) | SHAM Stimulation (N=6)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1) — A history of tinnitus for a participant was recorded at the start of the study. Symptoms worsened at 1 month follow up
Lightheadness (Nervous system disorders) | 0 (0) | 1 (1) — Lightheadedness experienced. Resolved on its own.

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed due to funding for a pilot study. There was a technical problem related to the NES task which resulted in the data not being collected after the first subject.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-13): https://cdn.clinicaltrials.gov/large-docs/54/NCT05165654/Prot_SAP_000.pdf